CLINICAL TRIAL: NCT06189833
Title: Phase 2 Study Applying Innovative Minimal Residual Disease (MRD) Techniques for Participants With Previously Untreated Multiple Myeloma Treated With D-VRd Prior To and After High-dose Therapy Followed by Autologous Stem Cell Transplantation (ASCT) - TAURUS
Brief Title: Phase 2 Study Applying MRD Techniques for Participants With Previously Untreated Multiple Myeloma Treated With D-VRd Prior To and After High-dose Therapy Followed by ASCT - TAURUS
Acronym: TAURUS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting European Myeloma Network (Network)
Collaborators: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Organization: European Myeloma Network B.V. (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMN33/54767414MMY2089
Record Dates: First submitted 2023-11-27; First posted 2024-01-05 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Multiple Myeloma
Keywords: MS-MRD
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Bortezomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- D-VRd + ASCT + DVRD (Experimental): Participants will receive daratumumab, bortezomib, lenalidomide and dexamethasone (DVRD) for 4 induction cycles prior to and 2 consolidation cycles following autologous stem cell transplantation.
  Daratumumab subcutaneously (SC), 1800 mg on days 1, 8, 15 and 22 of cycle 1 and 2, on days 1 and 15 of cycle 3-6 Bortezomib SC 1.3mg/m2 on days 1, 8, 15, 22 of cycle 1-6 Lenalidomide orally 25 mg once daily on days 1-21 of cycle 1-6 Dexamethasone 20 mg once daily on days 1, 2, 8, 9, 15, 16, 22 and 23 of cycle 1-6
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Daratumumab will be administered via a subcutaneous injection (SC)
  Other Names: JNJ-54767414
Drug: Bortezomib — Bortezomib will be administered via a subcutaneous injection (SC)
  Other Names: Velcade
Drug: Lenalidomide — Lenalidomide will be administered orally
Drug: Dexamethasone — Dexamethasone will be administered orally

SUMMARY:
This is a multicenter, single arm, open-label, Phase 2 study in mutiple myeloma with newly diagnosed and treatment-naïve participants for whom high-dose therapy and autologous stem cell transplantation is part of the intended treatment plan. The study is evaluating a technique called Mass Spectrometry Minimal Residual Disease (MS-MRD) using blood samples and compares it with the minimal residual disease (MRD) technique using bone marrow samples.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age, inclusive.
* Must have a new diagnosis of MM as per IMWG criteria.
* Measurable disease
* Newly diagnosed and treatment-naïve participants for whom high-dose therapy and autologous stem cell transplantation is part of the intended treatment plan.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
* Clinical laboratory values meeting the required criteria during screening and ≤3 days prior to receiving first study treatment dose.
* Adequate bone marrow function.
* Adequate liver function.
* Adequate renal function.
* A female of childbearing potential (FOCBP) must have two negative serum or urine pregnancy tests at screening including within 24 hours of the start of study treatment.
* Willing to practicing at least 1 highly effective method of contraception starting 4 weeks prior to start of study treatment, while receiving study treatment including during any dose interruptions, and for at least 3 months after the last dose of any component of the study treatment.

Exclusion Criteria:

* Prior or current systemic therapy or ASCT for any plasma cell dyscrasia, with the exception of emergency use of a short course (equivalent of dexamethasone 40 mg/day for a maximum 4 days) of corticosteroids before treatment.
* History of allogenic stem cell transplantation or prior organ transplant requiring immunosuppressive therapy.
* Peripheral neuropathy or neuropathic pain Grade 2 or higher, as defined by the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.
* Myelodysplastic syndrome or any malignancy within 24 months of signing consent. The only exceptions are malignancies treated within the last 24 months that are considered completely cured.
* Plasmapheresis ≤28 days of approval.
* Radiation therapy for treatment of plasmacytoma ≤14 days of approval of enrollment.
* Forced Expiratory Volume in 1 second (FEV1) <50% of predicted normal.
* Concurrent medical or psychiatric condition or disease.
* Myocardial infarction ≤6 months of enrollment, or an unstable or uncontrolled disease/condition related to or affecting cardiac function.
* Uncontrolled cardiac arrhythmia or clinically significant electrocardiogram (ECG) abnormalities.
* Allergy, hypersensitivity, or intolerance to boron or mannitol, corticosteroids, monoclonal antibodies or human proteins, or the excipients of daratumumab, lenalidomide, bortezomib or dexamethasone.
* Pregnant or breast-feeding females

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion (%) of agreement and disagreement in the MRD measurements in BM (by NGS-MRD) and in the MRD measurements in peripheral blood (by MS-MRD) at post-consolidation. | Up to 12 months
  The proportion (%) of agreement will be defined as the total number of concordant cases (i.e., MRD-positive by both techniques, MRD-negative by both techniques) versus the total number of cases with available results.

SECONDARY OUTCOMES:
Proportion (%) of agreement and disagreement in the MRD measurements in BM (by NGS-MRD) and in the MRD measurements in peripheral blood (by MS-MRD) at post-induction. | Up to 4 months and 2 weeks
  The proportion (%) of agreement will be defined as the total number of concordant cases (i.e., MRD-positive by both techniques, MRD-negative by both techniques) versus the total number of cases with available results.
Proportion (%) of agreement and disagreement in the MRD measurements in BM (by NGF-MRD) and in the MRD measurements in peripheral blood (by MS-MRD) at post-induction and post-consolidation. | Up to 12 months
  The proportion (%) of agreement will be defined as the total number of concordant cases (i.e., MRD-positive by both techniques, MRD-negative by both techniques) versus the total number of cases with available results.
Proportion (%) of agreement and disagreement in the MRD measurements in BM by NGF-MRD and NGS-MRD at post-induction and post-consolidation. | Up to 12 months
  The proportion (%) of agreement will be defined as the total number of concordant cases (i.e., MRD-positive by both techniques, MRD-negative by both techniques) versus the total number of cases with available results.
MRD negativity rate BM-MRD and PB-MRD | Up to 12 months
  To evaluate the MRD negativity rate achieved at any time up to the end of consolidation with BM based MRD techniques and with the MS-MRD technique
ORR, VGPR or better, CR or better, sCR at post-induction, post-transplant, post-consolidation and overall. | Up to 12 months
  ORR will be defined as the percentage of participants achieving confirmed PR or better (i.e., PR+VGPR+CR+sCR). The number and percentage of participants achieving ORR, VGPR or better, CR or better and sCR will be presented, post-induction, post-consolidation, post-transplant and overall.
Effect of cytogenetic abnormalities (presence or not), R-ISS (1, 2 or 3), CTCs (number of cells per ml) on likelihood to develop MRD-negative disease (with MS, NGS and NGF) and the agreement between the different techniques. | Up to 12 months
  Binary logistic regression will be used to identify factors associated with post-induction and post-consolidation MRD status (negative or positive) (as defined with NGS-MRD; NGF-MRD; MS-MRD; the most conservative method), in the MRD-evaluable Analysis Set. Odds ratios and respective 95% CIs will be estimated from univariable and multivariable models.

CONTACTS AND LOCATIONS:
Locations (31):
- Austria (4):
  - Innsbruck Medical University, Innsbruck
  - Ordensklinikum Linz, Linz
  - Clinic Ottakring, Vienna
  - Medical University of Vienna, Vienna
- Germany (2):
  - Universitätsklinikum Hamburg - Eppendorf, Hamburg
  - Klinikum rechts der Isar (MRI) der Technischen Universität München Department of Internal Medicine III (Hematology/Oncology) Munchen, München
- Greece (4):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - Alexandra General Hospital -Department of Clinical Therapeutics N.K. Univ. of Athens, Athens
  - St Savvas Cancer Hospital, Athens
  - Theagenion Cancer Hospital, Thessaloniki
- Italy (14):
  - AOU Ospedali Riuniti di Ancona, Ancona
  - ASST Papa Giovanni XXIII Hospital, Bergamo
  - A.O.U. di Bologna - Policlinico S. Orsola Malpighi, Bologna
  - A.O.Spedali Civili di Brescia, Brescia
  - A.O.U. Careggi - Firenze, Florence
  - A.O.U. Policlinico S. Martino - Ematologia, Genova
  - Novara Hospital, Novara
  - Policlinico S. Matteo Fondazione IRCCS - Pavia, Pavia
  - AUSL-IRCCS di Reggio Emilia Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale "Infermi" di Rimini, Rimini
  - Ematologia IRCCS Casa Sollievo della Sofferenza San Giovanni Rotondo, San Giovanni Rotondo
  - A.O. S. Santa Maria Hospital Institute of Oncohematology Terni, Terni
  - A.O.U. Città della Salute e della Scienza di Torino - SC Ematologia U, Torino
  - Ospedale S. Maria della Misericordia di Udine, Udine
- Netherlands (7):
  - Amsterdam Medical Center, Amsterdam
  - Rijnstate, Arnhem
  - Amphia ziekenhuis, Breda
  - University Medical Center Groningen, Groningen
  - Dijklander ziekenhuis, Purmerend
  - Erasmus University Medical Center Rotterdam, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam